CLINICAL TRIAL: NCT06391801
Title: Neuroathletic Training in Stroke Rehabilitation - A Pilot Study
Brief Title: Neuroathletic Training in Stroke Rehabilitation? A Single-blind Randomized Controlled Pilot Study on the Potentials of Neuroathletic Training on Balance Ability in Stroke Outpatient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Dr. Isabel Stolz, Research Associate, German Sport University, Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuroathletic in Stroke Rehab; 124/22 (Registry Identifier: Pilot study of specific neuroathletic training on the balance ability of stroke patients in outpatient rehabilitation)
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Balance Postural
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Daily 15 Minutes of Neuroathletic training additional to traditional movement therapy in outpatient rehabilitation
  Interventions: Behavioral: Neuroathletic training
- Control group (Active Comparator): Traditional movement therapy in outpatient rehabilitation
  Interventions: Behavioral: Traditional movement therapy in outpatient rehabilitation

INTERVENTIONS:
Behavioral: Neuroathletic training — Specific Neuroathletic training exercises were performed to improve balance ability of post stroke patients
  Arms: Intervention group
Behavioral: Traditional movement therapy in outpatient rehabilitation — Traditional movement therapy in outpatient rehabilitation
  Arms: Control group

SUMMARY:
Based on anecdotal evidence, neuroathletic training is described as effective for target groups in performance sports, leisure sports and movement therapy. Neuroathletic training is being integrated more and more into practical fields of training, coaching education and therapy. In addition to athletic objectives, it emphasizes to address central nervous system movement control and specific perception exercises, which are included in specific training sessions. It is gaining attention through literature and an increasing number of workshops for practitioners, yet scientific evidence to support effectiveness of therapeutic approaches is lacking. Only few research findings show positive effects in the context of specific neuroathletic exercises. With respect to patients in stroke rehabilitation, exercises to stimulate the visual and vestibular systems were found to be effective for movement rehabilitation. Exploring neuroathletic perceptual exercises to improve balance seems to be promising for the target group. Stroke patients experience deficits in balance and losses in motor function during activities of daily living, therefore temporal precision activity-related stimuli could provide a useful complement of movement therapy to provide targeted support of neuronal plasticity, in order to restore functions over time. Outpatient rehabilitation movement therapy aims to promote physical functions that are important in everyday life, including coordination and balance tasks, in order to enable independent and safe movement. To explore neuroathletic training potentials on balance ability in stroke rehabilitation, a single-blinded controlled pilot study was conducted in a stroke outpatient rehabilitation program.

DETAILED DESCRIPTION:
Study design The study design was a monocentric single-blinded randomized controlled pilot study (N=19). Aim of the study was to investigate potential effects of a 4-week outpatient rehabilitation program including 15 minutes of daily neuroathletic training compared to 15 minutes treatment as usual (traditional movement therapy). The primary endpoint was balance ability in stroke outpatient rehabilitation, measured via the German Version of the Berg Balance Scale (BBS) during a pre and post measurement, conducted by one blinded therapist in the years 2021-2022. The pretest of BBS was assessed in all participants on the first day of their rehabilitation program before the start of therapeutic measures. The second and final assessment of BBS was carried out on the last day after completion of all rehabilitation measures. Sample size calculation was based on an initial power analysis.

Population Participants were randomly assigned to the control and intervention groups by a coordinating therapist of the study site via a simple concealed randomization. Participant selection took place ad hoc. Inclusion criteria for the study participation were the main clinical diagnosis of stroke and indication for outpatient rehabilitation including movement therapy as well as adequate fitness to participate in a 4-week movement therapy program. All subjects agreed to participate voluntarily and gave written informed consent. The study was approved by Ethics Committee of the German Sports University Cologne in accordance with the Declaration of Helsinki (Seventh revision, 2013).

Study procedure The neuroathletic training included a structured exercise catalog prepared in advance and performed in a standardized manner for all patients of the intervention group. The conducting therapists received an introduction to carry out neuroathletic training and received all materials necessary for the intervention as well as the standardized training program with the exercise catalogue to perform almost identical training (table 1, Appendix A). All other therapeutic contents were the same for the intervention and control groups. More frequent short training sessions are to be preferred over a few longer ones. Therefore, training was conducted daily for 15 minutes with each patient. The total time of neuroathletic training in the intervention period was ten hours per patient of the intervention group.

Measures and statistical analyses As in the original English version, the German version of the Berg balance scale comprises 14 test items, which can be rated on a 5-point Likert scale from 0 to 4 points. It represents a well-established and valid measure and is considered as the gold standard to assess balance [12]. The total score is calculated by adding the values of each item and is a maximum of 56 points. According to Berg, Wood-Dauphinee, Williams & Maki [1992], persons with a total score of less than 45 points are considered to have impaired balance and are at increased risk of falling. The data analysis was carried out via IBM SPSS Statistics Version 28 (190). Demographic data were analyzed via descriptive statistics. The change in the subjects' ability to balance was analyzed in both groups using the Wilcoxon test. The examination of the values between the control and intervention group were analyzed using the Mann Whitney-U test (significance level α = 5 %) due to the small sample size. Effect sizes were calculated via Cohens d.

ELIGIBILITY:
Inclusion Criteria:

* main clinical diagnosis of stroke and indication for outpatient rehabilitation including movement therapy as well as adequate fitness to participate in a 4-week movement therapy program

Exclusion Criteria:

* No adequate fitness for participationg in the 4 week intervention time
* no adequate diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 4 weeks
  The BBS comprises 14 activities that the therapist observes and evaluates in relation to balance. A maximum of four points can be awarded for each activity.
  A maximum score of 56 points can be achieved. The therapist conducts the various activities according to an instructions (manual) and demonstrates them if necessary.
  Due to the very good reliability and responsiveness the scale can therefore be recommended for follow-up measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Oberberg - Healthcare facility, Gummersbach, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
The participants in this study did not give written consent for their personal data to be shared publicly; therefore, so due to the sensitive nature of the research, supporting data is unavailable.

REFERENCES:
- [Derived] Evers J, Stolz I, Klein M. Neuroathletic training in stroke rehabilitation? A single-blind randomized controlled pilot study on the potential of neuroathletic training for balance ability in stroke outpatient rehabilitation. BMC Res Notes. 2024 Dec 12;17(1):358. doi: 10.1186/s13104-024-07022-0. PMID 39668364